CLINICAL TRIAL: NCT01205932
Title: Randomized, Double-blind, Parallel-group, Active-controlled, Dose-confirmatory Bridging Study of Rivaroxaban (BAY59-7939) 5 to 10 mg Once-daily Regimen With a Reference Drug of Enoxaparin in the Prevention of Venous Thromboembolism in Patients Undergoing Elective Total Hip Replacement
Brief Title: Dose-confirmatory Bridging Study in Total Hip Replacement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 14397
Record Dates: First submitted 2010-09-19; First posted 2010-09-21 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Venous Thromboembolism
Keywords: venous thromboembolism; prevention; othopaedic surgery
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: Rivaroxaban (BAY59-7939)
- Arm 2 (Experimental)
  Interventions: Drug: Rivaroxaban (BAY59-7939)
- Arm 3 (Experimental)
  Interventions: Drug: Rivaroxaban (BAY59-7939)
- Arm 4 (Active Comparator)
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Rivaroxaban (BAY59-7939) — Daily dose: 5mg/day (5mg, once daily) for 34 to 35 days (±4 days)
  Arms: Arm 1
Drug: Rivaroxaban (BAY59-7939) — Daily dose: 7.5mg/day (7.5mg, once daily) for 34 to 35 days (±4 days)
  Arms: Arm 2
Drug: Rivaroxaban (BAY59-7939) — Daily dose: 10mg/day (10mg, once daily) for 34 to 35 days (±4 days)
  Arms: Arm 3
Drug: Enoxaparin — daily dose: 40mg/day (20mg each, twice daily) for 6 to 7 days (±2 days)
  Arms: Arm 4

SUMMARY:
The objective of this dose-confirmatory bridging study is to investigate the safety and efficacy of rivaroxaban 5 to 10 mg once-daily (od) dosing in the prevention of venous thromboembolism (VTE) in Japanese patients undergoing elective total hip replacement (THR) and to confirm the extrapolability of global data to Japanese patients by comparing with data from overseas phase II study (ODIXa-OD.HIP - Study 11527).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 20 years or above
* Patients undergoing elective THR (the first replacement of the applicable hip joint)
* Patients' written informed consent to participation after receiving detailed verbal and written information on any study specific procedures in advance

Exclusion Criteria:

* Planned, staged major orthopedic surgery within 3 months prior to elective THR or during this study
* History of clinically significant active bleeding (e.g. intracranial bleeding, gastrointestinal bleeding*), or high bleeding risk

  *: within 3 months prior to elective THR for gastrointestinal bleeding
* Subjects with hepatic disease which is associated with coagulopathy leading to a clinically relevant bleeding risk
* Severe impaired renal function (CLCR calculated by Cockcroft-Gault formula: <30 mL/min)
* Conditions prohibiting bilateral venography (e.g. amputation of 1 leg, allergy to contrast media)
* Ongoing anticoagulant therapy (e.g. warfarin, heparins and Factor Xa inhibitors other than study medication) that cannot be stopped (in the opinion of the investigator/sub investigator)
* Subjects for whom epidural catheters are expected to be left in for longer than 18 hours post-operatively
* Planned intermittent pneumatic compression during treatment period

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
A composite endpoint of any deep vein thrombosis (proximal and/or distal), non-fatal pulmonary embolism and death from all causes | Up to Day 9 (±2 days)
Treatment-emergent bleeding (major, non-major clinically relevant, other non-major) | Up to Day 8 (±2 days)

SECONDARY OUTCOMES:
Deep vein thrombosis (total, proximal, distal) | up to Day 9 (±2 days)
Symptomatic venous thromboembolism | up to Day 9 (±2 days)
Major venous thromboembolism (proximal deep vein thrombosis, pulmonary embolism or venous thromboembolism-related death) | up to Day 9 (±2 days)
Symptomatic venous thromboembolism | up to Day 36 (±4 days)
Symptomatic venous thromboembolism | within 30 days after stop of treatment with study drug.
Treatment-emergent bleeding (major, non-major clinically relevant, other non-major) | from the first intake of study medication to no later than 2 days after the last intake of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (35):
- Japan (35):
  - Nagoya, Aichi-ken
  - Matsudo, Chiba
  - Narashino, Chiba
  - Matsuyama, Ehime
  - Fukuoka, Fukuoka
  - Kōriyama, Fukushima
  - Asahikawa, Hokkaido
  - Hakodate, Hokkaido
  - Sapporo, Hokkaido
  - Kakogawa, Hyōgo
  - Kobe, Hyōgo
  - Nishinomiya, Hyōgo
  - Tsukuba, Ibaraki
  - Kagoshima, Kagoshima-ken
  - Kamakura, Kanagawa
  - Yokohama, Kanagawa
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Iida, Nagano
  - Sasebo, Nagasaki
  - Kurashiki, Okayama-ken
  - Tomigusuku, Okinawa
  - Hirakata, Osaka
  - Izumi, Osaka
  - Izumisano, Osaka
  - Kishiwada, Osaka
  - Osaka, Osaka
  - Sakai, Osaka
  - Sayama, Osaka
  - Suita, Osaka
  - Takatsuki, Osaka
  - Saga, Saga-ken
  - Nerima-ku, Tokyo
  - Setagaya City, Tokyo
  - Toyama, Toyama